CLINICAL TRIAL: NCT01093313
Title: Comparison of Attention Training and Cognitive Therapy in the Treatment of Social Phobia: a Randomized Controlled Trial
Brief Title: Attention Training and Cognitive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Dr Maree Abbott, The University of Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USydney9274
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Social Phobia
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention training (Experimental)
  Interventions: Behavioral: attention training
- Cognitive therapy (Active Comparator)
  Interventions: Behavioral: Cognitive therapy

INTERVENTIONS:
Behavioral: Cognitive therapy
  Arms: Cognitive therapy
Behavioral: attention training
  Arms: Attention training

SUMMARY:
The present study aimed to investigate the efficacy and process of change that occurs in Attention Training in comparison to an established treatment for social phobia, Cognitive Therapy. A randomized trial was conducted in which participants were allocated to either six weeks of Attention Training or Cognitive Therapy. It was hypothesized that both treatments would be effective in reducing social phobia symptoms, but that Attention Training would work primarily by reducing levels of self focused attention, while Cognitive Therapy would work through changes to probability and threat appraisals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age,
* be fluent in English
* have a primary concern of social anxiety that met DSM-IV criteria (APA, 2000) for social phobia. Both subtypes of social phobia, specific and generalized, were accepted into the study.

Exclusion Criteria:

* the presence of comorbid condition(s) that were more severe than the presenting social phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-08; Primary Completion 2007-04 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maree Abbott, PhD, Principal Investigator — University of Sydney
Locations (1):
- The University of Sydney, Sydney, New South Wales, Australia